CLINICAL TRIAL: NCT03222167
Title: Open-Label Multi-Center Single Arm Clinical Trial to Study the Efficacy and Safety of the Elbasvir/ Grazoprevir 50/100 mg Fixed Dose Combination Once Daily in Patients With Chronic HCV GT1b Infection Associated With Metabolic Syndrome
Brief Title: Open-Label Efficacy and Safety Study of the Elbasvir/ Grazoprevir Fixed Dose Combination Patients With Chronic HCV GT1b
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute Of Cardiology & Internal Diseases, Kazakhstan (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry); Synergy Research Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICID.HCV.0117
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-07

CONDITIONS: Chronic Hepatitis C Genotype 1B; Metabolic Syndrome; Fibrosis, Liver; Cirrhoses, Liver
Keywords: Elbasvir; Grazoprevir; SVR12; hepatitis C; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Liver Cirrhosis; Hepatitis C | interventions — elbasvir; grazoprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elbasvir/ Grazoprevir (Experimental): Elbasvir/ Grazoprevir 50/100 mg fixed dose combination for 12 weeks treatment aimed to evaluate SVR12 in treatment naïve patients with chronic hepatitis C (genotype 1b) infection, associated with metabolic syndrome, with or without severe fibrosis / compensated cirrhosis.
  Interventions: Drug: Elbasvir/ Grazoprevir 50/100 mg fixed dose combination

INTERVENTIONS:
Drug: Elbasvir/ Grazoprevir 50/100 mg fixed dose combination — Enrolled patients will be treated by Elbasvir/ Grazoprevir 50/100 mg fixed dose combination during 12 week. Followed-up on week 24. SVR12 will be evaluated.

SUMMARY:
This is a multi-center, open-label trial of Elbasvir/ Grazoprevir 50/100 mg fixed dose combination 12 week treatment aimed to evaluate SVR12 in treatment naïve patients with chronic hepatitis C (genotype 1b) infection, associated with of metabolic syndrome. The study to be conducted in conformance with Good Clinical Practices.

A total of 60 subjects will be studied at 2 sites in the Republic of Kazakhstan.

Males and Females treatment naïve patients with CHC genotype 1b infection associated with metabolic syndrome (MS), 18-70 years of age, with or without severe fibrosis / compensated cirrhosis will be enrolled. SVR 12 (primary endpoint) will be evaluated. Patients will be stratified by fibrosis stage and presence of metabolic syndrome components. Interim Analysis will be performed in order to estimate viral kinetics, applicability of SVR4 and durability of SVR12 by evaluation of virologic response at week 4 and 8 of treatment and follow-up at week 4 (SVR 4) and 24 will be performed - this will be a descriptive summary only without hypothesis testing.

The main hypothesis is that 12-week therapy with MK-5172 in combination with MK-8742 for treatment-naïve patients with HCV genotype 1b with metabolic syndrome is not notably worse than the same course for treatment-naïve patients with HCV genotype 1b without metabolic syndrome.

DETAILED DESCRIPTION:
60 treatment-naïve subjects with chronic hepatitis C genotype 1b infection associated with metabolic syndrome (MS), with or without severe fibrosis/compensated cirrhosis will be enrolled, males and females of 18-70 years of age.

Subjects will fulfill the following study visits: Day 1 (screening), Day 7, Week 2, Week 4, Week 8, Week 12, Week 24, Week 36.

Eligibility criteria re-checked, informed consent signed and medical history will be gathered on Day 1.

Treatment allocation and review study medication diary will be made on Day 7. Physical Examinations will be fulfilled on Day 1, Day 7, Week 4 and Week 12. Subject Confirmation of Birth Control and Review (Serious) Adverse Events will be made on every visit of subject.

Laboratory evaluations will include common blood analysis, urinalysis, biochemical blood analysis, Thyroid-stimulating hormone (TSH) and Т4 free, antigen testings (aHBs, HBsAg, HbeAg, aHDV, aHAV, aHEV, ANA, AMA, aHIV), HCV RNA (quantitative), HCV genotyping, Urine Pregnancy Test (females of child bearing potential only), Transient elastography, Calculation of APRI, Ultrasonography (of liver, gall bladder, spleen, pancreas), Upper GI Endoscopy.

Patients will be stratified by fibrosis stage and presence of metabolic syndrome components. Interim Analysis will be performed in order to estimate viral kinetics, applicability of SVR4 and durability of SVR12 by evaluation of virologic response at week 4 and 8 of treatment and follow-up at week 4 (SVR 4) and 24 will be performed - this will be a descriptive summary only without hypothesis testing.

Primary objectives:

• To demonstrate efficacy of 12 weeks therapy with MK-5172 (grazoprevir) in combination with MK-8742 (elbasvir) in treatment naïve patients with chronic hepatitis C (genotype 1b) with metabolic syndrome compared to patients without metabolic syndrome, as assessed by the proportion of subjects achieving SVR12, defined as HCV RNA < LLOQ (either TD[u] or TND) 12 weeks after the end of all study therapy.

Secondary objectives:

* To evaluate efficacy of 12 weeks therapy with MK-5172 in combination with MK-8742 in treatment naïve patients with chronic hepatitis C (genotype 1b) with metabolic syndrome compared to patients without metabolic syndrome, dependent on fibrosis stage, as assessed by the proportion of subjects achieving SVR12, defined as HCV RNA < LLOQ (either TD[u] or TND) 12 weeks after the end of all study therapy.
* To evaluate efficacy of MK-5172 in combination with MK-8742 in treatment naïve patients with chronic hepatitis C (genotype 1) combined with metabolic syndrome dependent on presence of the separate components of metabolic syndrome, as assessed by the proportion of subjects achieving SVR24, defined as HCV RNA < LLOQ (either TD[u] or TND) 12 weeks after the end of all study therapy.
* To evaluate efficacy of 12 weeks therapy with MK-5172 in combination with MK-8742 in treatment naïve patients with chronic hepatitis C (genotype 1b) with metabolic syndrome compared to patients without metabolic syndrome, as assessed by the proportion of TN subjects achieving undetectable (TND) HCV RNA and HCV RNA < LLOQ at Week 2, 4, 8 and Follow-Up Week 4 (SVR 4).
* To evaluate efficacy of 12 weeks therapy with MK-5172 in combination with MK-8742 in treatment naïve patients with chronic hepatitis C (genotype 1b) with metabolic syndrome compared to patients without metabolic syndrome, as assessed by the proportion of subjects achieving SVR24, defined as HCV RNA < LLOQ (either TD[u] or TND) 24 weeks after the end of all study therapy.
* To evaluate safety profile / adverse events of 12 weeks therapy with MK-5172 in combination with MK-8742 in treatment naïve patients with chronic hepatitis C (genotype 1b) with metabolic syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Be 18-70 years of age on a day of signing of informed consent.
2. Have ≤40 kg/m2.
3. Have HCV RNA ≥ 10,000 IU/mL at the time of screening.
4. Have documented chronic HCV GT1b (with no evidence of non-typeable or mixed genotype) infection (positive for anti-HCV antibody, HCV RNA, or HCV GT1b at least 6 months before screening).
5. Have liver disease staging assessment by means of liver biopsy performed within 12 calendar months prior to Day 1 of this study or Fibroscan performed within 6 calendar months prior to Day 1 of this study (cut-off of 12.5 kPa has a positive predictive value of 90% and a sensitivity of 95% for ≥F3).
6. Be HIV and HBV negative.
7. Be naïve to all anti-HCV treatment.
8. Have provided written informed consent for the trial.
9. Be diagnosed with metabolic syndrome (according to guidelines from the National Heart, Lung, and Blood Institute (NHLBI) and the American Heart Association (AHA)), i.e. have central obesity (defined as waist circumference in Asian males >94 cm, in Caucasian males >90 cm, in females > 80 cm) combined with at least any of two of the following factors: (1) raised triglycerides ≥150 mg/dL (1.7 mmol/L) or specific treatment for this lipid abnormality; (2) reduced HDL cholesterol < 40 mg/dL (1.03 mmol/L) in males or < 50 mg/dL (1.29 mmol/L) in females or specific treatment for this lipid abnormality; (3) raised blood pressure - systolic BP ≥130 or diastolic BP ≥ 85 mm Hg or treatment of previously diagnosed hypertension; (4) raised fasting plasma glucose (FPG) ≥100 mg/dL (5.6 mmol/L), or previously diagnosed type 2 diabetes.
10. Reproductive potential patient agrees to avoid becoming pregnant or impregnating a partner until at least 6 months after the last dose of medication.

Exclusion Criteria:

1. Is below 18 years of age.
2. Has not signed Informed Consent Document.
3. Has HCV genotype other than genotype 1b.
4. Has BMI > 40 kg/m2.
5. Has history of clinically significant psychiatric disorder which in the opinion of the investigator, would interfere with the study procedures and compliance.
6. Has received Peg/RBV, Telaprevir, or Boceprevir, or Sofosbuvir, or any other oral anti-HCV treatment/ combinations
7. Has documented portal hypertension and hepatic decompensation (Child-Pugh B or C, esophageal varices, ascites, elevated bilirubin, jaundice, splenomegaly, hepatic encephalopathy, albumin below 3 g/dl; platelet count < 75 000, INR<1.7), history of liver decompensation.
8. Has history of liver or other organ transplant.
9. Has autoimmune hepatitis.
10. Has ALT > 10 x ULN.
11. Is co-infected with hepatitis B virus (e.g., HBsAg positive) and HIV.
12. Has evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC (if liver imaging within 6 months of Day1 is not available, imaging is required during the screening).
13. Has a clinically-relevant drug or alcohol abuse within 12 months of screening.
14. Has decompensated DM with HbA1 >12%.
15. Has a medical/surgical condition that may result in a need for hospitalization during the period of the study.
16. Is a female who is pregnant or breast-feeding, or expecting to become pregnant and continue throughout treatment and follow up, OR male who plan to impregnate or has a female sexual partner of childbearing potential, or pregnant, or unwilling to commit to using a two methods of birth control throughout treatment and after the completion of all treatment and follow-up.
17. Is currently participating or has participated in a study with an investigational compound within 30 days
18. Is taking or plan to take any of the prohibited medications or herbal supplements: co-administration with the following drugs: Didanosine, Nafcillin, Rifampin Phenytoin, Bosentan, Modafinil, Phenobarbital, Carbamazepine, St. John's Wort (Hypericum perforatum), Glibenclamid, Glyburide, Gemfibrozil, Eltrombopag, Lapatinib, Efavirenz, Atazanavir, Darunavir, Lopinavir, Saquinavir, Tipranavir, Cyclosporine, Simvastatin, Fluvastatin, Rosuvastatin greater than 10 mg dose, Atorvastatine greater than 10 mg dose, hepatotoxic drugs. Any condition that requires administration of systemic corticosteroids, TNF antagonists, or other immunosuppressant drugs during the course of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
SVR12 evaluation | 12 weeks after the end of all study therapy (treatment success).
  The main outcome is SVR12, defined as HCV RNA < LLOQ (either TD[u] or TND)

SECONDARY OUTCOMES:
Death/Lost | 24 weeks
  Death or lost to follow-up before W24 will be considered as treatment failure (in full analysis set).

OTHER OUTCOMES:
HCV-RNA values | 24 weeks
  Definitively missing plasma HCV-RNA values at W24 will be considered as treatment failure

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Institute of Cardiology and Internal Medicine, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: No